CLINICAL TRIAL: NCT06172088
Title: Exploratory Study of Therapeutic Fasting to Reduce Limitations in Physical Well-being and Quality of Life During Endocrine Therapy With Aromatase Inhibitors
Brief Title: Exploratory Study Therapeutic Fasting Reduce Physical Limitations, Quality of Life During Aromatase Inhibitor Therapy
Acronym: FREE-AI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S00805-NIM
Record Dates: First submitted 2023-11-02; First posted 2023-12-15 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Patients Treated With Aromatase Inhibitors
Keywords: Fasting; Aromatase Inhibitors
MeSH Terms: conditions — Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Intervention Model Description: Bicenter, single-arm, prospective intervention study including qualitative accompanying study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therapeutic fasting for the reduction of physical of limitations in physical well-being and qol (Experimental)
  Interventions: Other: Fasting

INTERVENTIONS:
Other: Fasting — Sieben days of online supervised prolonged therapeutic fasting (max. 350 kcal/d).

SUMMARY:
In this explorative study, the feasibility of therapeutic fasting to reduce limitations in physical well-being and quality of life of patients undergoing endocrine therapy with aromatase inhibitors will be investigated. In addition, the application of the StudyU app, which is currently under development, will be monitored and the app adapted if necessary. In addition, in preparation for a larger multicenter main study, it will be examined whether the muscle and joint complaints frequently experienced by patients undergoing endocrine therapy with aromatase inhibitors (AI) can be alleviated by a 7-day guided therapeutic fasting intervention (prolonged fasting / PF) can be improved.

DETAILED DESCRIPTION:
After baseline (t0), all patients will receive the following intervention:

7 days of online supervised prolonged therapeutic fasting (max. 350 kcal/d).

Following the study intervention, at t1, patients will be offered a for a potential effect as sustainable as possible in addition to a dietary change.

According to the following criteria:

* As plant-based as possible
* Rich in nutritive prebiotics
* In addition, this group should include intermittent fasting/time restricted eating (16/8h) into their dietary habits (at least 6d/week).

All patients will be interviewed on a regular basis and anthropometric data will be collected accordingly at following time points:

* t1 (at the end of the fasting intervention).
* t2 (3 months after t0)

ELIGIBILITY:
Inclusion Criteria:

* Patients with curatively treated hormone receptor positive breast cancer who have been on aromatase inhibitors (AI) therapy for at least 3 months and have significant Pain (NRS>4).
* Informed consent.

Exclusion Criteria:

* Eating disorders.
* Permanent medication other than endocrine therapy, which would constitute an absolute or relative contraindication to outpatient fasting, such as Marcumar, lithium, Antiepileptic drugs, etc.
* Patients with diabetes mellitus type 1 or 2
* Uncontrolled cerebral seizure disorder.
* Participation in another diet/fasting study.
* Lack of willingness to store and share personal medical data within the framework of the protocol.
* Insufficient knowledge of the German language.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale | After 7 days (end of intervention)
  The numerical rating scale (NRS) will be used to assess the intensity of pain on a range of 0 to 10, with 0 as no pain and 10 as the most intense pain.
Brief Pain Inventory | After 7 days (end of intervention)
  The Brief Pain Inventory (BPI) scale will measure how pain has interfered with activities of daily living (general activity, walking, work, mood, enjoyment of life, relationships with others and sleep). Pain score: 1 - 4: Mild pain, 5 - 6: Moderate pain and 7 - 10: Severe pain.
Fibromyalgia Impact Questionnaire | After 7 days (end of intervention)
  The Fibromyalgia Impact Questionnaire (FIQ) has 10 items measuring physical functioning, mood, depression, anxiety, sleep, pain, stiffness, fatigue and well-being. Each item has a maximum score of 10 points, so the overall maximum score is 100.
Health Assessment Questionnaire-Diasbility Index | After 7 days (end of intervention)
  The Health Assessment Questionnaire-Diasbility Index (HAQ-DI) will be applied to assess the daily activity of patients, consists of 20 questions and is scored from 0 (no disability) to 3 (total disability).

SECONDARY OUTCOMES:
World Health Organization's 5 | After 7 days (end of intervention)
  The WHO-5 questionnaire will be used to assess the subjective mental well-being of patients. Each question is scored from 0 to 5. Low scores correspond to low level of well-being.
World Health Organization's 5 | Follow-up 3 Moths after the baseline.
  The WHO-5 questionnaire will be used to assess the subjective mental well-being of patients. Each question is scored from 0 to 5. Low scores correspond to low level of well-being.
Mindfulness and Awareness Scale | After 7 days (end of intervention)
  The Mindfulness and Awareness Scale (MAAS) measures a person's level of mindfulness in daily life. It evaluates how much time an individual spends in the present time. The scale ranges from 1 to 6 and consists of 15 items in total.
Mindfulness and Awareness Scale | Follow-up 3 Moths after the baseline.
  The Mindfulness and Awareness Scale (MAAS) measures a person's level of mindfulness in daily life. It evaluates how much time an individual spends in the present time. The scale ranges from 1 to 6 and consists of 15 items in total.
Relief of Cancer-related-Fatigue | After 7 days (end of intervention)
  The Relief of Cancer-related-Fatigue (BFI) is used to quickly assess the severity and impact of cancer-related fatigue. The questionnaire consists of 10 items covering six dimensions: Activity, mood, walking ability, work, relationship with others, and enjoyment of life. A score between 30 and 40 indicates moderate fatigue, scores above 70 indicate severe fatigue.
Relief of Cancer-related-Fatigue | Follow-up 3 Moths after the baseline.
  The Relief of Cancer-related-Fatigue (BFI) is used to quickly assess the severity and impact of cancer-related fatigue. The questionnaire consists of 10 items covering six dimensions: Activity, mood, walking ability, work, relationship with others, and enjoyment of life. A score between 30 and 40 indicates moderate fatigue, scores above 70 indicate severe fatigue.
Pittsburgh Sleep Quality Index | After 7 days (end of intervention)
  The Pittsburgh Sleep Quality Index (PSQI) measures subjective sleep quality. The questionnaire consists of 19 items and 7 component scores are obtained, each of which is scored from 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Pittsburgh Sleep Quality Index | Follow-up 3 Moths after the baseline.
  The Pittsburgh Sleep Quality Index (PSQI) measures subjective sleep quality. The questionnaire consists of 19 items and 7 component scores are obtained, each of which is scored from 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Blood pressure | After 7 days (end of intervention)
  It is defined as the force exerted by the blood on the arterial walls to circulate through the arteries and is measured in mm Hg. A normal value is considered to be less than 120/80 mmHg.
Blood pressure | Follow-up 3 Moths after the baseline.
  It is defined as the force exerted by the blood on the arterial walls to circulate through the arteries and is measured in mm Hg. A normal value is considered to be less than 120/80 mmHg.
Heart rate | After 7 days (end of intervention)
  It is defined as the number of times the heart pumps blood during a minute and is measured as the number of beats per minute. Between 60 and 100 beats per minute is considered a normal value.
Heart rate | Follow-up 3 Moths after the baseline.
  It is defined as the number of times the heart pumps blood during a minute and is measured as the number of beats per minute. Between 60 and 100 beats per minute is considered a normal value.
Food habits | Follow-up 3 Moths after the baseline.
  A standardized questionnaire will be used, where the following will be recorded: eating habits.
Body-Mass-Index | After 7 days (end of intervention)
  Body-Mass-Index (BMI) is a measure of body weight classification and is calculated based on weight and height, with the unit of measurement kg/m2. A BMI between 18.5 and 24.9 is considered normal weight, between 25 and 29.9 is defined as slightly overweight and a value above 30 is called severely overweight (obesity).
Body-Mass-Index | Follow-up 3 Moths after the baseline.
  Body-Mass-Index (BMI) is a measure of body weight classification and is calculated based on weight and height, with the unit of measurement kg/m2. A BMI between 18.5 and 24.9 is considered normal weight, between 25 and 29.9 is defined as slightly overweight and a value above 30 is called severely overweight (obesity).
Abdominal circumference | After 7 days (end of intervention)
  It is an anthropometric measurement used to establish the fat accumulated in a person in the abdominal area and is measured in centimeters (cm). For women, below 80cm is low risk, 80-88cm is high risk and more than 88cm is very high.
Abdominal circumference | Follow-up 3 Moths after the baseline.
  It is an anthropometric measurement used to establish the fat accumulated in a person in the abdominal area and is measured in centimeters (cm). For women, below 80cm is low risk, 80-88cm is high risk and more than 88cm is very high.
Triglycerides | After 7 days (end of intervention)
  Type of lipid found in the bloodstream and adipose tissue. Normal values are between 150-199 mg/dl, high between 200-499 mg/dl and very high values above 500 mg/dl.
Triglycerides | Follow-up 3 Moths after the baseline.
  Type of lipid found in the bloodstream and adipose tissue. Normal values are between 150-199 mg/dl, high between 200-499 mg/dl and very high values above 500 mg/dl.
Gamma-Glutamyl-Transferase | After 7 days (end of intervention).
  This is an enzyme found mainly in the liver. Its normal values are between 5-40 U/L.
Gamma-Glutamyl-Transferase | Follow-up 3 Moths after the baseline.
  This is an enzyme found mainly in the liver. Its normal values are between 5-40 U/L.
Fatty Liver Index | After 7 days (end of intervention)
  Fatty Liver Index (FLI) is a predictor of hepatic steatosis, calculated from BMI, waist circumference, y-GT and triglycerides.
Fatty Liver Index | Follow-up 3 Moths after the baseline.
  Fatty Liver Index (FLI) is a predictor of hepatic steatosis, calculated from BMI, waist circumference, y-GT and triglycerides.
Adverse events | After 7 days (end of intervention)
  Adverse events and serious adverse events are documented. Adverse events include any adverse symptoms, illnesses, disorders, or accidents that occur during the course of the study. Serious adverse events include events occurring during the course of the study that are immediately life-threatening and/or result in serious health problems (specifically, requiring unanticipated hospitalization or prolongation of hospitalization, or resulting in serious disability or incapacitation). The severity as well as the possible causal relationship with the intervention will be assessed by the study physician.
Adverse events | Follow-up 3 Moths after the baseline.
  Adverse events and serious adverse events are documented. Adverse events include any adverse symptoms, illnesses, disorders, or accidents that occur during the course of the study. Serious adverse events include events occurring during the course of the study that are immediately life-threatening and/or result in serious health problems (specifically, requiring unanticipated hospitalization or prolongation of hospitalization, or resulting in serious disability or incapacitation). The severity as well as the possible causal relationship with the intervention will be assessed by the study physician.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Loeffler, Dr, Principal Investigator — University Hospital Wuerzburg
Locations (2):
- Germany (2):
  - Robert-Bosch-Krankenhaus, Stuttgart, Baden Würtenberg
  - Würzburg University, Würzburg, Bavaria